CLINICAL TRIAL: NCT04268030
Title: High Order Spectral Analysis of Local Field Potential Data on a Subgroup of Parkinson's Disease Patients Who Are Carriers of Mutations in the Glucocerebrosidase (GBA) Gene Undergoing DBS Electrode Placement
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Gian Pal, Assistant Professor, Rush University Medical Center
Other Study IDs: 17112804-IRB02
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GBA mutation carriers with PD undergoing STN-DBS
  Interventions: Other: collection of LFPs

INTERVENTIONS:
Other: collection of LFPs — collection of local field potentials (LFPs) at rest and during hand opening and closing

SUMMARY:
The aim is to study a specific group of PD patients, carriers of mutations in the glucocerebrosidase (GBA) gene, which is the most common genetic risk factor for PD and is a harbinger of aggressive cognitive and motor decline. Approximately 12-17% of PD patients undergoing DBS are GBA mutation carriers. GBA mutation carriers with PD have a specific phenotype characterized by more significant motor dysfunction and reduced short-term visual memory function compared with their non-GBA counterparts. Thus as GBA mutation carriers have a "signature" phenotype, the investigators hypothesize that these GBA mutation carriers have a unique "signature" of oscillatory activity that can be distinguished from non-mutation carriers during motor activation and during cognitive tasks. Identification of this "signature" will provide critical information that is required to: 1) understand the underlying neurophysiological mechanisms responsible for the aggressive disease course of GBA associated PD, and 2) further develop customized adaptive DBS systems.

ELIGIBILITY:
Inclusion Criteria:

* undergoing bilateral STN-DBS
* diagnosis of Parkinson's disease

Exclusion Criteria:

* no Parkinson's disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease (PD) with and without mutations in the GBA gene who already have an implanted deep brain stimulator (DBS) device or those patients with PD-GBA mutation carrier who will be undergoing placement of a DBS device using standard technique with sedation and local anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
change in beta symmetry | 1 day
  LFP

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No